CLINICAL TRIAL: NCT04297709
Title: Study of Urinary Predictors of Exacerbations by Biomarkers in Cystic Fibrosis (SUPERB-CF)
Brief Title: Study of Urinary Predictors of Exacerbations by Biomarkers in Cystic Fibrosis
Acronym: SUPERB-CF
Status: Completed | Type: Observational
Sponsor: Mologic Ltd (Industry)
Collaborators: Heart of England NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: SUPERB-CF
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study of Urinary Predictors of Exacerbations by Biomarkers in Cystic Fibrosis

DETAILED DESCRIPTION:
People with cystic fibrosis (CF) are prone to chest infections (pulmonary exacerbations) and suffer premature death due to respiratory failure. Patients that experience more frequent pulmonary exacerbations have worse prognosis and early antibiotic treatment of pulmonary exacerbations is therefore one of the major goals of CF care. Antibiotic treatment is often currently delayed, since we rely on patients contacting the CF team when they develop worsening symptoms. We hypothesise that if we could allow patients to detect and receive treatment for early pulmonary exacerbations by measuring urinary biomarkers, this would minimise lung damage and result in improved clinical outcomes.

In phase 1, 40 patients will be asked to collect daily urine samples, in addition to recording daily spirometry and a daily symptom score for 4 months. Phase 1 aims to identify the urinary biomarkers that are associated with CF pulmonary exacerbations. In phase 2, the same 40 patients will be asked to collect and test a daily urine sample using a novel testing device in addition to recording daily spirometry and a daily symptom score for 4 months. Phase 2 aims to validate the use of the urine testing device as a method of diagnosing early pulmonary exacerbations.

In summary, this study aims to develop and validate a novel noninvasive point of care (near-patient) diagnostic testing system, to allow people with CF to diagnose early pulmonary exacerbations by measuring urinary biomarkers. If successful, we hope that this will provide patients with an easy to use device, which will empower patients and their caregivers to treat exacerbations at an earlier stage, with potential health and economic benefits.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed CF diagnosis
* Aged >18 years of age
* Patients able and willing to give informed consent
* Requirement for at least one course of intravenous antibiotics for a pulmonary exacerbation within the previous 3 months.

Exclusion Criteria:

* Patients not able or not willing to give informed consent
* Patients who are currently participating in another clinical trial (excluding observational studies)
* Pneumothorax or lung surgery within the previous 3 months, eye surgery (e.g. cataract operation) in the previous 4 weeks, or any other factor that prevents safe measurement of spirometry.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with CF
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Measurement of biomarkers in the urine of CF patients to assess their potential for predicting exacerbations | 4 months
  Signalling molecules/acute phase proteins e.g. Interleukin 6 (IL-6), Interleukin 8 (IL-8), N-Formyl methionine Leucyl phenylalanine (fMLP), Fibrinogen, C-reactive protein (CRP).
  Proteases & proteolytic activity, e.g. Matrix metalloproteases (MMP's), Myeloperoxidase (MPO), Human neutrophil elastase (HNE), Cathepsins.
  Protease inhibitors, e.g. Tissue inhibitor of Metalloproteinase (TIMP), Alpha-1 anti-Trypsin (A1AT), Cystatin C, Secretory leukocyte peptidase inhibitor (SLPI).
  Degradation products e.g. Desmosine and Elastin Fragments, Acetyl PGP (Ac-PGP).
  Metabolites and other urinary markers, e.g. Creatinine, Human Serum Albumin (HSA), Retinol Binding Protein 4 (RBP4), Beta 2 Microglobulin (B2M).
  Other markers of interest, e.g. Siglec 8, Chitinase 3 like 1 protein, Club cell protein 16 (CC16).
  Note. Concentrations of all these biomarkers are expressed in microgramme/ml

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Nash, BSc, Principal Investigator — Heart of England NHS Foundation Trust
Locations (1):
- Birmingham Heartlands Hospital, Birmingham, United Kingdom